CLINICAL TRIAL: NCT01235728
Title: A Double Blind, Active-Comparator-, and Vehicle-Controlled, Multiple-Dose Study to Evaluate the Efficacy and Pharmacokinetics of MK-0873 in Patients With Plaque Psoriasis
Brief Title: A Study to Evaluate and Compare the Efficacy and Pharmacokinetics of MK-0873 for the Treatment of Plaque Psoriasis (MK-0873-022)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 0873-022
Record Dates: First submitted 2010-11-04; First posted 2010-11-05 (Estimated); Results first posted 2014-06-11 (Estimated); Last update posted 2019-02-08 (Actual); Status verified 2019-01

CONDITIONS: Psoriasis; Plaque Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — MK 0873

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (8):
- Treatment Sequence 1 (Experimental): Participants were randomized to receive MK-0873 on upper lesion A and vehicle on upper lesion B, and MK-0873 on lower lesion C and calcitriol on lower lesion D.
  Interventions: Drug: MK-0873 2% Cream; Drug: MK-0873 vehicle (placebo) Cream; Drug: Calcitriol Cream
- Treatment Sequence 2 (Experimental): Participants were randomized to received MK-0873 on lower lesion A and vehicle on lower lesion B, and MK-0873 on upper lesion C and calcitriol on upper lesion D.
  Interventions: Drug: MK-0873 2% Cream; Drug: MK-0873 vehicle (placebo) Cream; Drug: Calcitriol Cream
- Treatment Sequence 3 (Experimental): Participants were randomized to receive MK-0873 on upper lesion A and vehicle on upper lesion B, and calcitriol on lower lesion C and MK-0873 on lower lesion D.
  Interventions: Drug: MK-0873 2% Cream; Drug: MK-0873 vehicle (placebo) Cream; Drug: Calcitriol Cream
- Treatment Sequence 4 (Experimental): Participants were randomized to receive MK-0873 on lower lesion A and vehicle on lower lesion B, and calcitriol on upper lesion C and MK-0873 on upper lesion D.
  Interventions: Drug: MK-0873 2% Cream; Drug: MK-0873 vehicle (placebo) Cream; Drug: Calcitriol Cream
- Treatment Sequence 5 (Experimental): Participants were randomized to receive vehicle on upper lesion A and MK-0873 on upper lesion B, and MK-0873 on lower lesion C and calcitriol on lower lesion D.
  Interventions: Drug: MK-0873 2% Cream; Drug: MK-0873 vehicle (placebo) Cream; Drug: Calcitriol Cream
- Treatment Sequence 6 (Experimental): Participants were randomized to receive vehicle on lower lesion A and MK-0873 on lower lesion B, and MK-0873 on upper lesion C and calcitriol on upper lesion D.
  Interventions: Drug: MK-0873 2% Cream; Drug: MK-0873 vehicle (placebo) Cream; Drug: Calcitriol Cream
- Treatment Sequence 7 (Experimental): Participants were randomized to receive vehicle on upper lesion A and MK-0873 on upper lesion B, and calcitriol on lower lesion C and MK-0873 on lower lesion D.
  Interventions: Drug: MK-0873 2% Cream; Drug: MK-0873 vehicle (placebo) Cream; Drug: Calcitriol Cream
- Treatment Sequence 8 (Experimental): Participants were randomized to receive vehicle on lower lesion A and MK-0873 on lower lesion B, and calcitriol on upper lesion C and MK-0873 on upper lesion D.
  Interventions: Drug: MK-0873 2% Cream; Drug: MK-0873 vehicle (placebo) Cream; Drug: Calcitriol Cream

INTERVENTIONS:
Drug: MK-0873 2% Cream — Approximately 3 to 5 mg of MK-0873 2% cream per cm^2 of body area in 2 divided applications per day for 28 days. The maximum area for one treatment will be approximately 5% of body surface area.
Drug: MK-0873 vehicle (placebo) Cream — Approximately 3 to 5 mg matching placebo to MK-0873 2% cream per cm^2 of body area in 2 divided applications per day for 28 days. The maximum area for one treatment will be approximately 5% of body surface area.
Drug: Calcitriol Cream — Approximately 3 to 5 mg of Calcitriol 0.0003% (3 µg/g) per cm^2 of body area once daily for 28 days. The maximum area for one treatment will be approximately 5% of body surface area

SUMMARY:
This is a within-participant comparison study to investigate the efficacy of a 28-day regimen of MK-0873 2% cream twice a day (b.i.d.) compared to MK-0873 vehicle (matching placebo) b.i.d. as well as to a positive control comparator calcitriol 0.0003% (3 µg/g) in participants with plaque psoriasis. In order to be enrolled in the study, patients need to have at least two pairs (lesions AB and CD) of approximately similar plaque lesions in severity and size of surface area involved and located in approximately symmetric regions such as the trunk or limbs of the body. Participants will be randomly assigned to apply either MK-0873 or MK-0873 vehicle to plaque A or B and will be randomly assigned to apply MK-0873 or calcitriol to plaque C or D. It is hypothesized that MK-0873 cream formulation administered to participants with psoriasis by the topical route will result in a statistically greater percent target lesion severity (TLS) reduction in plaque lesion than will MK-0873 Vehicle on Day 29.

ELIGIBILITY:
Inclusion Criteria

* Is a male or female 18 to 65 years of age
* Female subjects of reproductive potential must have a negative serum pregnancy test at screening and agree to use and/or have their partner use two (2) acceptable methods of birth control
* Has a Body Mass Index (BMI) ≤36 kg/m^2 (up to 40 kg/m^2 may be enrolled, in consultation with Sponsor)
* Has diagnosis of plaque-type psoriasis at least 6 month prior to administration of study drug (participants with concurrent psoriatic arthritis may be enrolled)
* Has plaque-type psoriasis with at least two pairs of symmetrically located plaque lesions that exhibit similar baseline TLS values (TLS in each plaque ≥6 and

  ± 2 points difference between left and right plaque lesions)
* Has plaque-type psoriasis with lesion severity score ≥4 covering at least 1 to 20% of total body surface area at screening and at baseline.
* Is judged to be in good health based on medical history, physical examination, vital sign measurements, electrocardiogram assessment, and laboratory safety tests

Exclusion Criteria

* Has nonplaque forms of psoriasis (e.g., Erythrodermic, guttate, or pustular).
* Has current drug-induced psoriasis (e.g., a new onset of psoriasis or an exacerbation of psoriasis from beta blockers, calcium channel blockers or lithium).
* Has received phototherapy or any systemic medications/treatments that could affect psoriasis or TLS evaluation (including but not limited to oral or injectable corticosteroids, retinoids, 1, 25-dihydroxy vitamin D3 and analogues, psoralens, sulfsalazine, hydroxyurea, fumaric acid derivatives, or herbal treatments) within 4 weeks of study drug administration.
* Has used topical medications/treatments that could affect psoriasis or TLS evaluation (e.g., corticosteroids, coal tar, anthralin, calcipotriene, topical vitamin D derivatives, retinoids, tazarotene, methoxsalen, trimethyl psoralens) within 2 weeks of study drug administration.
* Has used any systemic immunosuppressants (e.g., Methotrexate, azathioprine, cyclosporine, 6-thioguanine, mercaptopurine, mycophenolate mofetil, hydroxyurea, or tacrolimus) within 4 weeks of study drug administration or biologics (e.g., anti-tumor necrosis factor [TNF], anti-interleukins) within 3 months of study drug administration.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-11-01 (Actual); Primary Completion 2011-04-01 (Actual); Study Completion 2011-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (2):
- United States (2):
  - Call for Information, Fort Myers, Florida
  - Call for Information, Miramar, Florida

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=0873-022&kw=0873-022&tab=access

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Sequence 2: Participants were randomized to receive MK-0873 on lower lesion A and vehicle on lower lesion B, and MK-0873 on upper lesion C and calcitriol on upper lesion D.
- Treatment Sequence 4: Participants were randomized to receive MK-0873 on lower lesion A and vehicle on lower lesion B, and calcitriol on upper lesion C and MK-873 on upper lesion D.
Period: Overall Study
Arm/Group | Treatment Sequence 1 | Treatment Sequence 2 | Treatment Sequence 3 | Treatment Sequence 4 | Treatment Sequence 5 | Treatment Sequence 6 | Treatment Sequence 7 | Treatment Sequence 8
Started | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 2 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- MK-0873: Participants were randomized to receive MK-0873 on upper or lower lesion C or D and calcitriol on the opposing lesion D or C. The lesion receiving calcitriol was evaluated.
Arm/Group | MK-0873
Number analyzed (Participants) | 24
Age, Continuous [Mean (Full Range); unit: Years] | 43.3 [30 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 17

OUTCOME MEASURES:

1. Primary Outcome: Least Squares Mean Percent Change From Baseline (Predose Day 1) of Target Lesion Severity (TLS) Score for Lesions Treated With MK-0873 and Lesions Treated With MK-0873 Vehicle
Description: Each lesion was evaluated for 3 components: erythema, induration, and scaling. Each component was given a score using the following scale: 0=none, 1=slight, 2=moderate, 3=marked, 4=very marked, with increasing score reflecting increased lesion severity. The TLS score (range 0 to 12) is calculated as the sum of the 3 components.
Time Frame: Baseline and Day 29
Population: The population consisted of all participants that received treatment, had no major protocol violations, and had TLS scores available at baseline and Day 29.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Units Other Than Participants: Lesions
Groups:
- MK-0873: Participants were randomized to receive MK-0873 on upper or lower lesion C or D and calcitriol on the opposing lesion D or C. The lesion receiving MK-0873 was evaluated.
- MK-0873 Vehicle: Participants were randomized to receive MK-0873 vehicle on upper or lower lesion A or B and MK-0873 on the opposing lesion B or A. The lesion receiving MK-0873 vehicle was evaluated.
Arm/Group | MK-0873 | MK-0873 Vehicle
Number analyzed (Participants) | 23 | 23
Number analyzed (Lesions) | 23 | 23
Percent Change | -47.37 [-56.87 to -37.86] | -42.71 [-52.21 to -33.22]

2. Secondary Outcome: Least Squares Mean Percent Change From Baseline (Predose Day 1) of TLS Score for Lesions Treated With MK-0873 and Lesions Treated With Calcitriol
Description: as for outcome 1
Time Frame: Baseline and Day 29
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Units Other Than Participants: Lesions
Groups:
- Calcitriol 0.0003%: Participants were randomly assigned to receive calcitriol 0.0003% (3mg/g) BID for 28 days on upper or lower lesion C or D and MK-0873 on the opposing lesion D or C. The lesion receiving calcitriol was evaluated.
Arm/Group | Calcitriol 0.0003% | MK-0873
Number analyzed (Participants) | 23 | 23
Number analyzed (Lesions) | 23 | 23
Percent Change | -57.24 [-66.82 to -47.67] | -47.89 [-57.39 to -38.40]

3. Secondary Outcome: Mean Maximum Plasma Concentrations at Trough of Day 8, 15, 22, and 29 Following Topical Administration of MK-0873 to Psoriatic Patients
Description: Plasma samples were collected at 12 hours post-dose on Days 8, 15, 22, and 28 to evaluate the mean maximum plasma concentration at trough of MK-0873.
Time Frame: Day 8, 15, 22, 29
Population: The population consisted of all participants that received treatment, had no major protocol violations, and had MK-0873 plasma trough values available for the Day 8, 15, 22, and 28 treatment.
Measure: Mean (Standard Deviation); unit: nM
Groups:
- MK-0873: Participants were randomized to receive MK- 0873 on upper or lower lesion A or B and MK-0873 Vehicle on the opposing lesion B or A, and MK-0873 on upper or lower lesion C or D and calcitriol on the opposing lesion D or C.
Arm/Group | MK-0873
Number analyzed (Participants) | 23
nM | 3.6 (3.1)

ADVERSE EVENTS:
Arm/Group | MK-0873
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 8/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-0873 (N=24)
Nasopharyngitis (Infections and infestations) | 3 (3)
Headache (Nervous system disorders) | 3 (3)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation.